CLINICAL TRIAL: NCT05394285
Title: A Multicenter, Randomized, Self-controlled Exploratory Clinical Study of Hetrombopag Olamine Tablets for Thrombocytopenia Induced by Anti-tumor Treatment in Advanced Breast Cancer
Brief Title: A Clinical Study of Hetrombopag Olamine Tablets for Thrombocytopenia Induced by Anti-tumor Treatment in Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNCH-MBC10
Record Dates: First submitted 2022-04-30; First posted 2022-05-27 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — hetrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hetrombopag Olamine tablets (Experimental): The first anti-tumor treatment cycle (multicenter, open label, randomized controlled):
  When platelets were <50*109/L, oral hetrombopag 7.5 mg/day was started. When the platelet count is >100*109/L, the administration is suspended.
  2nd anti-tumor treatment cycle (exploratory study): Prophylactic use (60 cases in the test group and the control group): oral hetrombopag 7.5 mg/day (initial dose) was started on d2 after anti-tumor treatment for 14 days.
  Interventions: Drug: Hetrombopag
- rhTPO (Other): The first anti-tumor treatment cycle (multicenter, open label, randomized controlled):
  Start using rh-TPO 15000 units/day (subcutaneous injection) when platelets are less than 50*109/L. When the platelet count is more than 100*109/L, the administration is suspended.
  2nd anti-tumor treatment cycle (exploratory study): Prophylactic use (60 cases in the test group and the control group): oral hetrombopag 7.5 mg/day (initial dose) was started on d2 after anti-tumor treatment for 14 days.
  Interventions: Drug: Hetrombopag

INTERVENTIONS:
Drug: Hetrombopag — The first anti-tumor treatment cycle (multicenter, open label, randomized controlled):
  When platelets were <50*109/L, oral hetrombopag 7.5 mg/day was started. When the platelet count is >100*109/L, the administration is suspended.
  2nd anti-tumor treatment cycle (exploratory study): Prophylactic use (60 cases in the test group and the control group): oral hetrombopag 7.5 mg/day (initial dose) was started on d2 after anti-tumor treatment for 14 days.

SUMMARY:
This study now plans to explore the efficacy and safety of hetrombopag in cancer therapy-induced thrombocytopenia in advanced breast cancer, so as to further guide the clinical application of hetrombopag in chemotherapy-induced platelets.

DETAILED DESCRIPTION:
Cancer therapy-induced thrombocytopenia increases the risk of hemorrhagic complications, the need for platelet transfusions, and limits the dose of cytotoxic drugs in the treatment of certain malignancies. Thrombopoietin receptor agonist (TPO-RA) has a therapeutic effect on cancer therapy-induced thrombocytopenia (CTIT). As an innovative TPO-RA drug, hetrombopag has a more optimized molecular structure and reduced liver and kidney toxicity. A registrational Phase III clinical study in CTIT patients is ongoing. This study now plans to explore the efficacy and safety of hetrombopag in cancer therapy-induced thrombocytopenia in advanced breast cancer, so as to further guide the clinical application of hetrombopag in therapy-induced platelets.

ELIGIBILITY:
Inclusion Criteria:

1. The patients signed the informed consent and voluntarily joined the study;
2. Age 18-75 years old, male or female;
3. Patients with advanced breast cancer diagnosed by histopathology or cytology, who are receiving and continue to receive the same chemotherapy regimen;
4. Can accept the current chemotherapy regimen (must be platinum-containing chemotherapy regimen: lobaplatin, carboplatin, cisplatin, etc.) for at least 2 cycles;
5. The first occurrence of platelets <50×109/L in the current chemotherapy cycle;
6. The investigator determines that the patient can receive hetrombopag administration;
7. Neutrophil count ≥ 1.0×109/L, hemoglobin ≥ 80g/L before administration of Haitrombopag;
8. Life expectancy at screening ≥ 12 weeks;
9. ECOG: 0-1;
10. The main organ functions are normal, and there are no serious complications.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding;
2. Unable to understand the research nature of the research or have not obtained informed consent;
3. The investigator judges other circumstances that are not suitable for inclusion in the study;
4. Thrombocytopenia caused by other causes (chronic liver disease, sepsis, disseminated intravascular coagulation, immune thrombocytopenia, etc.);
5. Patients with unstable angina pectoris, congestive heart failure, uncontrolled hypertension, uncontrolled arrhythmia or recent history (within 1 year of screening) of myocardial infarction;
6. Those with a history of blood disease or tumor bone marrow infiltration;
7. Those who received simultaneous radiotherapy and those who received pelvic radiotherapy in the past;
8. Arterial or venous thrombotic events within the past 6 months;
9. There are currently uncontrollable infections;
10. Clinical manifestations of severe bleeding within 2 weeks before screening, such as gastrointestinal or central nervous system bleeding;
11. Need emergency treatment, such as superior vena cava syndrome, spinal cord compression;
12. The absolute value of neutrophils is less than 1.0×109/L, and the hemoglobin is less than 80g/L, and granulocyte colony-stimulating factor, red blood cells, and EPO infusion therapy in accordance with clinical routine are allowed;
13. Obvious abnormal liver function: patients without liver metastases, ALT/AST>3ULN (upper limit of normal value), TBIL>3ULN; patients with liver metastases, ALT/AST≥5ULN, TBIL≥5ULN;
14. Abnormal renal function: serum creatinine ≥ 1.5ULN or eGFR ≤ 60 ml/min (Cockcroft-Gault formula);

16. Received thrombopoietin receptor agonist drugs (such as Eltrombopag, Romigrastim), or recombinant human thrombopoietin (rhTPO), recombinant human interleukin-11 (rhIL) within 1 month before screening -11) Treatment; 17. Received platelet transfusion within 3 days before randomization; 18. Patients with known or expected hypersensitivity or intolerance to the active ingredients or excipients of Hetrombopag ethanolamine tablets.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The response rates to platelet-raising therapy in prevention stage | 30day±3day after the last administration of Hetrombopag Olamine Tablets
  The response rate defined as the proportion of pts not requiring platelet transfusion or adjustment (dose reduction 20%, treatment delays for ≥5 days, or treatment discontinuation) due to thrombocytopenia, and not developing severe thrombocytopenia (PLT < 25×10⁹/L, or PLT <50×10⁹/L for >7 days).

SECONDARY OUTCOMES:
The response rate to platelet-raising therapy in treatment stage; | 30day±3day after the last administration of Hetrombopag Olamine Tablets or rh TPO
  The response rate defined as the treatment of pts not requiring platelet transfusion or adjustment (dose reduction 20%, treatment delays for ≥5 days, or treatment discontinuation) due to thrombocytopenia, and not developing severe thrombocytopenia (PLT < 25×10⁹/L, or PLT <50×10⁹/L for >7 days).
The lowest platelet value after anti-tumor treatment; | 30day±3day after the last administration of Hetrombopag Olamine Tablets
  The lowest platelet value after anti-tumor treatment;
The incidence of platelets <50×109/L and <25×109/L; | 30day±3day after the last administration of Hetrombopag Olamine Tablets
  The incidence of platelets <50×109/L and <25×109/L;
The duration of platelets <50×109/L and <25×109/L; | 30day±3day after the last administration of Hetrombopag Olamine Tablets
  The duration of platelets <50×109/L and <25×109/L;
The time for platelets to recover to more than 100×109/L; | 30day±3day after the last administration of Hetrombopag Olamine Tablets
  The time for platelets to recover to more than 100×109/L;
latelet recovery to the highest value after anti-tumor treatment; | 30day±3day after the last administration of Hetrombopag Olamine Tablets
  latelet recovery to the highest value after anti-tumor treatment;
the incidence of adverse events; | 30day±3day after the last administration of Hetrombopag Olamine Tablets
  the incidence of adverse events;

CONTACTS AND LOCATIONS:
Overall Officials: min yan, Principal Investigator — Henan Cancer Hospital
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No